CLINICAL TRIAL: NCT03499860
Title: Prediction of Fluid Responsiveness From Passive Leg Raising Induced Changes in Perfusion Index and Pleth Variability Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mountain Emergency Medicine (Other)
Collaborators: Department of Anaesthesiology, Merano Hospital, Italy (Unknown)
Responsible Party: Principal Investigator, Simon Rauch, Researcher, Institute of Mountain Emergency Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 06
Record Dates: First submitted 2018-03-31; First posted 2018-04-17 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Fluid Responsiveness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Passive Leg Raising Test — A passive leg raising test is performed in all patients included in the study

SUMMARY:
The aim of the study is to evaluate whether changes in Perfusion Index (PI) and Pleth Variability Index (PVI) during passive leg raising test can predict fluid responsiveness in spontaneously breathing patients.

Fluid responsive patients are defined as showing an increase in cardiac output >10% during a passive leg raising test, measured semi-invaseively with FloTrac® (Edwards LifeSciences. Irvine, United States).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the intensive or intermediate care unit after abdominal surgery (including urological and gynecological surgery performed in laparotomy)
* Spontaneous breathing
* Arterial line already in place
* Oral and written informed consent obtained

Exclusion Criteria:

* Age <18 years
* Abdominal trauma as the reason for surgery
* Missing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
PI difference | 90 seconds
  Difference in the change of perfusion index from baseline during a passive leg raising maneuver in fluid responsive patients compared to fluid non-responders
PVI difference | 90 seconds
  Difference in the change of pleth variability index from baseline during a passive leg raising maneuver in fluid responsive patients compared to fluid non-responders

CONTACTS AND LOCATIONS:
Locations (1):
- "F. Tappeiner" Hospital Merano, Merano, Bolzano, Italy